CLINICAL TRIAL: NCT04313322
Title: Treatment of COVID-19 Patients Using Wharton's Jelly-Mesenchymal Stem Cells
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Stem Cells Arabia (Other)
Responsible Party: Principal Investigator, Adeeb Al Zoubi, President, Chief Scientific Officer, Stem Cells Arabia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: COVID-19
Record Dates: First submitted 2020-03-15; First posted 2020-03-18 (Actual); Last update posted 2020-03-18 (Actual); Status verified 2020-03

CONDITIONS: Use of Stem Cells for COVID-19 Treatment
Keywords: Stem Cells, COVID-19, SARS CoV2, WJ MSCs, Immunomodulation,
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: Patients positively diagnosed with COVID-19
Masking Description: None. This is a direct study for the potential effects of WJ-MSCs on COVID-19 outcome.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- WJ-MSCs (Experimental): WJ-MSCs will be derived from cord tissue of newborns, screened for HIV1/2, HBV, HCV, CMV, Mycoplasma, and cultured to enrich for MSCs.
  WJ-MSCs will be counted and suspended in 25 ml of Saline solution containing 0.5% human serum Albumin, and will be given to patient intravenously.
  Interventions: Biological: WJ-MSCs

INTERVENTIONS:
Biological: WJ-MSCs — WJ-MSCs will be derived from cord tissue of newborns, screened for HIV1/2, HBV, HCV, CMV, Mycoplasma, and cultured to enrich for MSCs.
  WJ-MSCs will be counted and suspended in 25 ml of Saline solution containing 0.5% human serum Albumin, and will be given to patient intravenously.

SUMMARY:
The purpose of this study is to investigate the potential use of Wharton's Jelly Mesenchymal stem cells (WJ-MSCs) for treatment of patient diagnosed with Corona Virus SARS-CoV-2 infection, and showing symptoms of COVID-19.

DETAILED DESCRIPTION:
COVID-19 is a condition caused by infection with Coronoa Virus (SARS-CoV-2). This virus has a high transmission rate and is spreading at very high rates. causing a worldwide pandemic. Patients diagnosed with COVID-19 and confirmed positive with the virus, will be given three IV doses of WJ-MSCs consisting of 1X10e6/kg. The three doses will be 3 days apart form each other.

Patients will be followed up for a period of three weeks to assess the severity of the condition and measure the viral titers.

ELIGIBILITY:
Inclusion Criteria:

COVID-19 positive according to diagnosis and clinical management of COVID-19 criteria.

Exclusion Criteria:

* Participants in other clinical trials
* patients with malignant tumors
* pregnant and lactating women
* co-infection with other infectious viruses or bacteria
* History of several allergies
* Patients with history of pulmonary embolism
* any liver or kidney diseases
* HIV positive patients
* Considered by researchers to be not suitable to participate in this clinical trial
* Chronic heart failure with ejection fraction less than 30%.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2020-03-16 (Estimated); Primary Completion 2020-06-30 (Estimated); Study Completion 2020-09-30 (Estimated)

PRIMARY OUTCOMES:
Clinical outcome | 3 weeks
  Improvement of clinical symptoms including duration of fever, respiratory destress, pneumonia, cough, sneezing, diarrhea.
CT Scan | 3 weeks
  Side effects measured by Chest Readiograph
RT-PCR results | 3 weeks
  Results of Real-Time Polymerase Chain Reaction of Viral RNA, Turing negative

SECONDARY OUTCOMES:
RT-PCR results | 8 weeks
  Results of Real-Time Polymerase Chain Reaction of Viral RNA, Turing negative

CONTACTS AND LOCATIONS:
Locations (1):
- Stem Cells Arabia, Amman, Jordan

IPD SHARING:
Plan to Share IPD: No